CLINICAL TRIAL: NCT05101395
Title: Prevalence of H. Pylori Gastritis in Sleeve Gastrectomy Specimens: A Cross-Sectional
Brief Title: Prevalence of H. Pylori Gastritis in Sleeve Gastrectomy Specimens
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Ibrahim Mansour, Senior General Surgery Resident, University of Jordan
Other Study IDs: 10/2020/8972
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Gastritis H Pylori; Gastritis; Obesity Associated Disorder
Keywords: Histopathology; Sleeve gastrectomy; LSG; Gastritis; H. Pylori; Jordan; Middle East
MeSH Terms: conditions — Gastritis | interventions — Azure Stains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Gastritis: Patients who underwent sleeve gastrectomy and the histopathology result of resected gastric specimen showed the presence of gastritis in it.
  Interventions: Other: Giemsa stain

INTERVENTIONS:
Other: Giemsa stain — Giemsa special stain was employed for detection of H. Pylori microorganisms.

SUMMARY:
This is a cross-sectional study looking for prevalence of H.Pylori related gastritis among patients underwent sleeve gastrectomy over five year study period. The study also looks for possible association with patients's characteristics. Also, compares its findings with similar regional and international studies.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent sleeve gastrectomy
* surgery was performed between January 2015 and October 2019

Exclusion Criteria:

* patients whose resected specimens were not examined histopathologically

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Obese patients who undergo sleeve gastrectomy for bariatric reasons
Sampling Method: Probability Sample
Enrollment: 810 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of gastritis | start to end of the study, 5 years
  proportion of patients who underwent sleeve gastrectomy who have gastritis in their resected gastric specimen at or during study period.
  calculated as (number of pt with gastritis / number of examined resected gastric specimens)
Prevalence of H.pylori gastritis | start to end of the study, 5 years
  proportion of patients who underwent sleeve gastrectomy who have H.pylori related gastritis in their resected gastric specimen at or during study period.
  calculated as (number of pt with H.pylori gastritis / number of examined resected gastric specimens)

SECONDARY OUTCOMES:
Prevalence of other histopathological findings | start to end of the study, 5 years
  proportion of patients who underwent sleeve gastrectomy who have histopathological findings not including gastritis or H.pylori related gastritis in their resected gastric specimen at or during study period.
  calculated as (number of pt with the histopathological finding / number of examined resected gastric specimens)
likelihood ratio between H.pylori gastritis and advancing age | start to end of the study, 5 years
  The relationship between H.pylori gastritis and advancing age. likelihood ratio will be calculated by cross table analysis using Statistical Analysis Software SPSS program version 26.
likelihood ratio between H.pylori gastritis and female gender | start to end of the study, 5 years
  The relationship between H.pylori gastritis and female gender. likelihood ratio will be calculated by cross table analysis using Statistical Analysis Software SPSS program version 26.
likelihood ratio between H.pylori gastritis and BMI | start to end of the study, 5 years
  The relationship between H.pylori gastritis and body mass index (BMI). weight and height will be combined to report BMI in kg/m^2 likelihood ratio will be calculated by cross table analysis looking for using Statistical Analysis Software SPSS program version 26.

CONTACTS AND LOCATIONS:
Overall Officials: Raed Al-Taher, M.D., Study Director — Jordan University Hospital; Mohammad Z Rashdan, M.D., Principal Investigator — Jordan University Hospital; Firas I Obeidat, Prof., Study Chair — Jordan University Hospital
Locations (1):
- Jordan University Hospital, Amman, Jubaiha, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
We are not willing to share study data due to hospital policies, but data is available for interested researchers upon request after verification and masking through corresponding author.

REFERENCES:
- [Background] Boliko MC. FAO and the Situation of Food Security and Nutrition in the World. J Nutr Sci Vitaminol (Tokyo). 2019;65(Supplement):S4-S8. doi: 10.3177/jnsv.65.S4. PMID 31619643
- [Background] Ge L, Moon RC, Nguyen H, de Quadros LG, Teixeira AF, Jawad MA. Pathologic findings of the removed stomach during sleeve gastrectomy. Surg Endosc. 2019 Dec;33(12):4003-4007. doi: 10.1007/s00464-019-06689-y. Epub 2019 Feb 15. PMID 30771070
- [Background] Rosenthal RJ; International Sleeve Gastrectomy Expert Panel; Diaz AA, Arvidsson D, Baker RS, Basso N, Bellanger D, Boza C, El Mourad H, France M, Gagner M, Galvao-Neto M, Higa KD, Himpens J, Hutchinson CM, Jacobs M, Jorgensen JO, Jossart G, Lakdawala M, Nguyen NT, Nocca D, Prager G, Pomp A, Ramos AC, Rosenthal RJ, Shah S, Vix M, Wittgrove A, Zundel N. International Sleeve Gastrectomy Expert Panel Consensus Statement: best practice guidelines based on experience of >12,000 cases. Surg Obes Relat Dis. 2012 Jan-Feb;8(1):8-19. doi: 10.1016/j.soard.2011.10.019. Epub 2011 Nov 10. PMID 22248433
- [Background] Abd Ellatif ME, Abdallah E, Askar W, Thabet W, Aboushady M, Abbas AE, El Hadidi A, Elezaby AF, Salama AF, Dawoud IE, Moatamed A, Wahby M. Long term predictors of success after laparoscopic sleeve gastrectomy. Int J Surg. 2014;12(5):504-8. doi: 10.1016/j.ijsu.2014.02.008. Epub 2014 Feb 18. PMID 24560848
- [Background] Safaan T, Bashah M, El Ansari W, Karam M. Histopathological Changes in Laparoscopic Sleeve Gastrectomy Specimens: Prevalence, Risk Factors, and Value of Routine Histopathologic Examination. Obes Surg. 2017 Jul;27(7):1741-1749. doi: 10.1007/s11695-016-2525-1. PMID 28063114
- [Background] Yardimci E, Bozkurt S, Baskoy L, Bektasoglu HK, Gecer MO, Yigman S, Akbulut H, Coskun H. Rare Entities of Histopathological Findings in 755 Sleeve Gastrectomy Cases: a Synopsis of Preoperative Endoscopy Findings and Histological Evaluation of the Specimen. Obes Surg. 2018 May;28(5):1289-1295. doi: 10.1007/s11695-017-3014-x. PMID 29151240
- [Background] Miller GC, Reid AS, Brown IS. The pathological findings seen in laparoscopic sleeve gastrectomies for weight loss. Pathology. 2016 Apr;48(3):228-32. doi: 10.1016/j.pathol.2015.12.449. Epub 2016 Mar 8. PMID 27020497
- [Background] F. Obeidat, A. Shahait, H. Shanti, H. Al-Momani, and S. Abu Halaweh, "Histopathology results of Jordanian patients after laparoscopic sleeve gastrectomy," Saudi J. Obes., vol. 3, no. 1, p. 18, 2015, doi: 10.4103/2347-2618.158693
- [Background] Deitel M, Gagner M, Erickson AL, Crosby RD. Third International Summit: Current status of sleeve gastrectomy. Surg Obes Relat Dis. 2011 Nov-Dec;7(6):749-59. doi: 10.1016/j.soard.2011.07.017. Epub 2011 Aug 10. PMID 21945699
- [Background] Agha R, Abdall-Razak A, Crossley E, Dowlut N, Iosifidis C, Mathew G; STROCSS Group. STROCSS 2019 Guideline: Strengthening the reporting of cohort studies in surgery. Int J Surg. 2019 Dec;72:156-165. doi: 10.1016/j.ijsu.2019.11.002. Epub 2019 Nov 6. PMID 31704426
- [Background] Buchwald H, Oien DM. Metabolic/bariatric surgery worldwide 2011. Obes Surg. 2013 Apr;23(4):427-36. doi: 10.1007/s11695-012-0864-0. PMID 23338049
- [Background] Angrisani L, Santonicola A, Iovino P, Formisano G, Buchwald H, Scopinaro N. Bariatric Surgery Worldwide 2013. Obes Surg. 2015 Oct;25(10):1822-32. doi: 10.1007/s11695-015-1657-z. PMID 25835983
- [Background] Angrisani L, Santonicola A, Iovino P, Vitiello A, Zundel N, Buchwald H, Scopinaro N. Bariatric Surgery and Endoluminal Procedures: IFSO Worldwide Survey 2014. Obes Surg. 2017 Sep;27(9):2279-2289. doi: 10.1007/s11695-017-2666-x. PMID 28405878
- [Background] B. A. Hussein, A. Khammas, J. Anglo, A. Al Mazrouei, and F. Badri, "Is Histopathology Needed after Sleeve Gastrectomy?," J. Am. Coll. Surg., vol. 227, no. 4, p. e71, 2018, doi: 10.1016/j.jamcollsurg.2018.08.192
- [Background] Al Saady R, Ejeckam G. Histopathological findings in laparoscopic sleeve gastrectomy specimens. Qatar Med J. 2019 Jul 25;2019(1):5. doi: 10.5339/qmj.2019.5. eCollection 2019. PMID 31384574
- [Background] S. R. Shikha Jain, "Histopathological Spectrum of Laparoscopic Sleeve Gastrectomies: A Retrospective Study," Indian J Pathol Res Pr., vol. 8, no. 2, pp. 223-228, 2019, doi: http://dx.doi.org/10.21088/ijprp.2278.148X.8219.16.